CLINICAL TRIAL: NCT07162038
Title: Phase I Trial Integrating HLA-Haploidentical Anti-CD19 CAR T Cells With Post-Transplantation Cyclophosphamide-Based HLA-Haploidentical Hematopoietic Cell Transplantation
Brief Title: Phase I Trial Integrating HLA-Haploidentical Anti-CD19 CAR-T Cells With Post-Transplantation Cyclophosphamide-Based HLA-Haploidentical Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001785; 001785-C
Record Dates: First submitted 2025-09-06; First posted 2025-09-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Hematologic Malignancies; Hematologic Neoplasms
Keywords: Chimeric-Antigen-Receptor T-cell Therapy; High Risk Hematologic Malignancy; CD19; Hematopoietic Cell Transplant
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Cyclophosphamide; Mycophenolic Acid; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Donor (No Intervention): Donors for Arms 1 and 2
- Phase I: Dose Escalation (Experimental): Participants receiving CAR-T cells at escalation/de-escalation dose levels to determine MTD
  Interventions: Biological: mCD19-CAR-CD28-CD3-zeta.(anti-CD19 CAR) retroviral vector-transduced allogeneic peripheral blood lymphocytes (PBL); Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Sirolimus; Device: CD19 Flow Cytometry Assay; Device: CD19 Immunohistochemical Assay; Radiation: Total Body Irradiation
- Phase I: Dose Expansion (Experimental): Participants receiving CAR-T cells at MTD
  Interventions: Biological: mCD19-CAR-CD28-CD3-zeta.(anti-CD19 CAR) retroviral vector-transduced allogeneic peripheral blood lymphocytes (PBL); Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mycophenolate Mofetil; Drug: Sirolimus; Device: CD19 Flow Cytometry Assay; Device: CD19 Immunohistochemical Assay; Radiation: Total Body Irradiation

INTERVENTIONS:
Biological: mCD19-CAR-CD28-CD3-zeta.(anti-CD19 CAR) retroviral vector-transduced allogeneic peripheral blood lymphocytes (PBL) — CAR-T cell infusion given at four escalating dose levels (DL1: 3 x 10^4 cells/kg, DL2: 1 x 10^5 cells/kg, DL3: 3 x 10^5 cells/kg, DL4: 1 x 10^6 cells/kg) with a dose de-escalation dose (DL-1: 1 x 10^4 cells/kg), if needed.
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion
Drug: Fludarabine — Pre-transplant: 30 mg/m^2 IV infusion over 30-60 minutes once daily for 5 days from day -6 through day -2
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion
Drug: Cyclophosphamide — Pre-transplant: 14.5 mg/kg/day IV daily for 2 days pre-transplant on day -6 and day -5.
  Post-transplant: 25 mg/kg/day on day +3 and day +4.
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion
Drug: Mycophenolate Mofetil — 15 mg/kg orally or IV three times daily (max 1000 mg/dose) starting on day +5, continued through day +35 post-transplant.
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion
Drug: Sirolimus — Loading dose of 6 mg orally given on day +5, then maintenance dose starting at 2 mg orally daily on day +6 with dose adjustments to maintain a trough of 5-12 ng/ml, continued through day +60 post-transplant.
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion
Device: CD19 Flow Cytometry Assay — Assay used to determine CD19+ status
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion
Device: CD19 Immunohistochemical Assay — Assay used to determine CD19+ status
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion
Radiation: Total Body Irradiation — 400 centigray (cGy) to be delivered in 2 fractions as 200 cGy per fraction twice a day on Day -1 pre-transplant.
  Arms: Phase I: Dose Escalation; Phase I: Dose Expansion

SUMMARY:
Background:

High-risk blood cancers (leukemias and lymphomas) often come back after treatment, and many cannot be cured with chemotherapy alone. These cancers may be treated and potentially cured in 2 ways: (1) Bone marrow transplant (allogeneic hematopoietic cell transplantation, or alloHCT) gives immune and blood stem cells from a donor. These new cells can attack the cancer and also grow into healthy blood. (2) Chimeric antigen receptor (CAR) T-cell therapy takes immune cells and changes them in a lab to better recognize and target certain cancers. But these 2 treatments are not usually given at the same time.

Objective:

To test alloHCT and CAR-T cell therapy, used together, in people with high-risk blood cancers.

Eligibility:

People aged 18 to 75 years with an aggressive blood cancer that has a protein on the surface called CD19. A healthy related donor aged 12 years or older is also needed; this donor may be a parent or child or may be some siblings or even extended family members, but has to be half-matched at something called the HLA (human leukocyte antigen).

Design:

Participants will be screened. They will have imaging scans, blood tests, and tests of their heart and lung function. They will have eye and dental exams. They may have fluid drawn from around their spinal cord (spinal tap) and tissue taken from inside a bone (bone marrow biopsy).

Healthy donors will provide bone marrow, immune cells, and about 9 tablespoons of blood for both the recipient s treatment and for research. They will also provide stool, saliva, and oral swabs just for research.

Recipient participants will stay in the hospital for 4 to 6 weeks. They will be given drugs over 6 days to prepare for the cell therapies. Both the donor bone marrow cells and CAR-T-cells will be given through a tube inserted into a vein. They will receive drugs to reduce complications after the treatments.

Participants will remain within a 1-hour drive of the hospital for 2 to 3 months after they leave the hospital. They will have frequent visits during that time. They will continue to have periodic follow-up visits for 5 years.

...

DETAILED DESCRIPTION:
Background:

* High-risk hematologic malignancies generally are incurable without an allogeneic hematopoietic cell transplant (HCT), but even with HCT they are at high-risk of relapse and poor overall survival.
* Chimeric-antigen-receptor (CAR) T-cell therapy can offer a high remission rate for relapsed or refractory B-cell malignancies but is not curative in the majority of patients.
* Currently, these two therapies (HCT and CAR-T cells) are used individually or sequentially, with HCT being used as consolidation or salvage post-CAR-T cells or CART cells being used to treat post-HCT relapse.
* Allogeneic CAR-T cells may be given to treat post-transplant relapse, but have not been used early post-transplant due to potential increased risk of graft-versus-host disease (GVHD).
* Post-transplantation cyclophosphamide (PTCy) reduces rates of severe acute and chronic GVHD and the immunosuppressive burden after HCT, including allowing LAhaploidentical HCT to be performed safely and routinely worldwide.
* In pre-clinical major histocompatibility complex (MHC)-haploidentical HCT models, CAR-T cells can be given on day 0 or day +5 (before or early after PTCy) and exert potent anti-tumor effects without impairing PTCy s efficacy in preventing GVHD. Administration of CAR-T cells on day +9 or +14 was ineffective in eradicating leukemia.
* In our preclinical models, administration of CAR-T cells on day 0 (prior to PTCy) surprisingly led to better anti-tumor efficacy than when given on day +5, associated with better early expansion, less CD4+ CAR-T cells with a regulatory phenotype, more activated CD4+ CAR-T cells, and more cytotoxic CD8+ CAR-T cells.
* The premise for the clinical application is that the CAR-T cells given in conjunction with or early post-transplant would induce an initial deep remission, while the polyclonal allogeneic T cells contained in the HCT would eliminate escape clones and promote longterm cure.
* The direct integration of CAR-T cells with PTCy-based HCT has the potential to provide synergistic reduction of relapse, reduce the duration of treatment, and allow CAR-T cells to persist post-transplant.

Objectives:

* To identify the safety of donor-derived HLA-haploidentical anti-CD19 CAR-T cells that can be given in combination with PTCy-based HLA-haploidentical allogeneic HCT in participants who have high-risk CD19-expressing hematologic malignancies (Phase I -dose escalation).
* To estimate 1 year relapse and survival outcomes at the maximum tolerated dose (MTD) (Phase I - dose expansion)

Eligibility:

* Adults age 18-75 years
* High-risk CD19-expressing hematologic malignancies
* Available HLA-haploidentical donor
* Adequate organ function
* KPS >= 60%

Design:

* Open-label, single-center, non-randomized, phase I study
* All recipient participants will receive reduced intensity conditioning, HLA-haploidentical bone marrow HCT, GVHD prophylaxis including post-transplantation cyclophosphamide, and allogeneic donor-derived anti-CD19 CAR-T cells.
* The study will proceed to a small, four-level phase I dose escalation study based on the standard 3+3 approach. CAR-T cells will be administered on day 0, except in the case of dose de-escalation wherein alternative dose levels would be employed and CAR-T cells would then be administered on day +7.
* Dose-escalation will be based on absence of grade III-IV acute GVHD (aGVHD), severe cytokine release syndrome (CRS), severe neurotoxicity or other toxicities as specified, or non-relapse mortality by day +28
* We will expand to include 6 additional participants at the maximum tolerated dose level determined by the phase I dose escalation to better estimate relapse and GVHD outcomes. Recipient participants will be followed for 5 years.

ELIGIBILITY:
-INCLUSION CRITERIA - Recipient

1. Participants with high or very high-risk hematologic malignancies, as defined by the revised Disease Risk Index (DRI), or malignancy that remains persistently MRD+ (by flow cytometry, cytogenetics, FISH, PCR, or NGS) on most recently assessed disease specimen (within 2 months of initiating conditioning).
2. Hematologic malignancy must be CD19+ (uniform expression on immunohistochemistry or >= 80% on flow cytometry) as confirmed by CD19 IHC assay (BT51E) or flow cytometry (BD QuantiBRITE(TM) Beads PE Fluorescence Quantitation Kit). (Participants do not have to have refused or lack access to commercial anti-CD19 CAR-T-cell therapies since this study focuses on the integration of CAR-T cells and HCT and not specifically the CAR-T cells themselves; furthermore the construct used to manufacture this product is the same as used in a current commercial product, but developed from a new batch and with a similar but not identical manufacturing process.)
3. Age 18-75
4. Karnofsky >= 60%.
5. Participants must have adequate organ and marrow function as defined below:

   * Cardiac ejection fraction >= 45% by 2D echocardiography;
   * Forced expiratory volume-1 (FEV-1) and diffusing capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) all of >= 50% predicted;
   * Estimated serum creatinine clearance of >= 60 ml/minute/1.73m^2 calculated using eGFR in the clinical lab (participants with estimated serum creatinine clearance less than 60 may have measured creatinine clearance performed and if >= 60 will be considered eligible);
   * Total bilirubin <= 2X the upper limit of normal (participants with documented or suspected Gilbert s are exempt from this requirement);
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 5X the upper limit of normal.
6. At least one available HLA-haploidentical donor
7. Women of child-bearing potential (WOCBP) must agree to use a highly effective method of contraception (hormonal, intrauterine device (IUD), surgical sterilization, abstinence) at the study entry and for 1 year after transplant (restriction period).

   Men must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) at the study entry and for 1 year after transplant. We also will recommend men with female partners of childbearing potential to ask female partners to be on highly effective birth control (hormonal, intrauterine device (IUD), surgical sterilization). Men must not freeze or donate sperm within the same period.
8. Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 1 year after transplant.
9. Participants seropositive for human immunodeficiency virus (HIV) not due to intravenous immunoglobulin, must have been on effective combination anti-retroviral therapy for 6 months and without detectable viral load prior to the beginning of conditioning.
10. For participants seropositive for hepatitis B virus (HBV) core antibody not due to intravenous immunoglobulin, a HBV viral load should be undetectable.
11. Participants seropositive for hepatitis C virus (HCV) not due to intravenous immunoglobulin must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
12. Ability of participant to understand and the willingness to sign a written informed consent document.
13. Ability and willingness of participant to co-enroll on 20-C-0051: Gene Therapy Follow Up Protocol for Subjects Previously Enrolled in NCI for Immuno-Oncology Studies

14 Willingness to remain in the NIH hospital or, if discharged, stay close to the NIH (<60 minutes drive), for a minimum of 100 days after transplant or longer if there are complications. Participants must commit to having an adult caregiver with them during the first 100 days after transplant in case of discharging from the hospital before 100 days.

INCLUSION CRITERIA - Donor

1. Related donor (age >=12) deemed suitable, eligible, and willing to donate, per clinical evaluations, who are additionally willing to donate blood, bone marrow, and stool for research. Related donors will be evaluated in accordance with existing Standard Policies and Procedures for determination of eligibility and suitability for clinical donation.

EXCLUSION CRITERIA - Recipient

1. Participants who are receiving any other investigational agents within 3 weeks prior to the beginning of conditioning.
2. Active CNS involvement of primary hematologic malignancy
3. Active malignancy of non-hematopoietic type (excluding non-melanoma skin cancers) which is metastatic, relapsed/refractory to treatment, or locally advanced and not amenable to intended curative treatment per standard of care.
4. Prior checkpoint inhibitor therapy within 6 weeks prior to the beginning of conditioning.
5. Prior history of seizure.
6. Uncontrolled infection.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents used in study.
8. Positive beta-HCG serum or urine pregnancy test performed in females of childbearing potential at screening. (A low positive test in a post-menopausal woman may not be exclusionary if deemed not indicative of pregnancy per gynecology.)
9. Uncontrolled intercurrent illness evaluated by medical history, physical exam, EKG, and laboratory testing (e.g., severe endocrinopathy, disseminated intravascular coagulation, profound electrolyte disturbance) that would make it unsafe to proceed with transplantation.

EXCLUSION CRITERIA - donor

1. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Identify the safety of anti-CD19 CAR T-cell therapy in combination with HLA-haploidentical HCT in participants with high risk CD19+ hematologic malignancies | 28 days (or 35 days for alternate dose levels)
  Determine the fraction of evaluable recipient participants at each dose level who experience a dose-limiting toxicity (DLT).
Estimate the 1 year relapse and survival outcomes at the maximum tolerated dose | 1 year
  Estimates will be determined using Kaplan-Meier curves or competing risk-based cumulative incidence curves as appropriate for participants treated at the MTD and may be reported individually for the MTD and other dose levels. The results at indicated time points will be reported and may include 95% confidence intervals as appropriate.

SECONDARY OUTCOMES:
Estimate the incidence and severity of CRS and ICANS | 100 days
  Rate and grade of CRS and ICANS will be measured by the maximum grade as assessed by the ASTCT Consensus Criteria for each condition and reported as fractions of those that attained each grade of severity.
Estimate the incidence of Grade II-IV and Grade III-IV acute GVHD at +200 days | 200 days
  Grade II-IV and III-IV aGVHD will be evaluated descriptively including fractions who attain each condition, along with 95% confidence intervals as appropriate.
Estimate the incidence and severity of chronic GVHD at 1 year | 1 year
  Analyses will be done numerically and using cumulative incidence curves with 95% confidence intervals at the stated time points as appropriate.
Estimate incidence of primary engraftment failure and kinetics of engraftment | 60 days
  Will be reported as a proportion of evaluation participants
Estimate relapse/progression, non-relapse mortality, progression-free survival, and overall survival at 1 year | 1 year
  Analyses will be done numerically and using cumulative incidence curves with 95% confidence intervals at the stated time points as appropriate.
Estimate relapse/progression, non-relapse mortality, progression-free survival, and overall survival at 5 years | 1 year
  Analyses will be done numerically and using cumulative incidence curves with 95% confidence intervals at the stated time points as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001785-C.html